CLINICAL TRIAL: NCT01224145
Title: A Phase II, Single-dose, Open-label Study to Investigate the Feasibility and Efficacy of the CollaRx® Bupivacaine Implant (200 mg Bupivacaine Hydrochloride) in Men After Laparoscopic Inguinal or Umbilical Herniorrhaphy
Brief Title: Assess the Feasibility and Efficacy of the CollaRx® Bupivacaine Implant Laparoscopic Inguinal or Umbilical Herniorrhaphy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INN-CB-011
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Hernia; Postoperative Pain
MeSH Terms: conditions — Hernia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: laparoscope for bupivacaine sponge (200 mg bupivacaine hydrochloride) placement in laparoscopic hernia repair.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: Bupivacaine Collagen Sponge (Experimental): bupivacaine collagen sponges
  Interventions: Drug: 5x5cm bupivacaine collagen sponges

INTERVENTIONS:
Drug: 5x5cm bupivacaine collagen sponges
  Other Names: Bupivacaine collagen implant

SUMMARY:
This study will assess pain intensity for the first 72 hrs after aggravated movement (cough) following Laparoscopic Inguinal or Umbilical Herniorrhaphy.

DETAILED DESCRIPTION:
Inguinal herniorrhaphy is a common surgery; approximately 2,800 per million people in the United States (US) undergo the procedure annually.Common surgical methods of herniorrhaphy include open and laparoscopic placement of synthetic mesh. Studies have shown that the use of synthetic mesh greatly reduces the risk of hernia recurrence regardless of the method used for its placement. Furthermore, utilizing the laparoscopic approach for umbilical hernia repair, specifically with the use of mesh, may also reduce the risk of infection.

Bupivacaine is a local anesthetic (pain medicine) that has an established safety profile. Collagen is a protein that is found in all mammals. The CollaRx Bupivacaine implant is a thin flat sponge made out of collagen that comes from cow tendons and contains bupivacaine. When inserted into a surgical site, the collagen breaks down and bupivacaine is released at the site but very little is absorbed into the blood stream. The high levels of bupivacaine at the surgical site may result in less pain for several days after surgery.

This open-label study will assess pain intensity after surgery in patients who receive the CollaRx Bupivacaine implant as well as determine the feasibility of the use of the laparoscope for sponge placement in laparoscopic hernia repair.

ELIGIBILITY:
Inclusion Criteria:

1. Man ≥18 years
2. Has a planned unilateral inguinal herniorrhaphy (laparoscopy, transabdominal preperitoneal [TAPP] approach or totally extraperitoneal [TEP] approach) or laparoscopic umbilical herniorrhaphy to be performed according to standard surgical technique under general anesthesia.
3. Willing to use opioid rescue analgesia.

Exclusion Criteria:

1. Has a known hypersensitivity to amide local anesthetics, opioids, or bovine products.
2. Scheduled for bilateral inguinal herniorrhaphy.
3. Undergone a prior herniorrhaphy at the location scheduled for repair.
4. Undergone major surgery within 3 months of the scheduled herniorrhaphy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03-22 (Actual); Primary Completion 2011-06-20 (Actual); Study Completion 2011-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (1):
- Research Concepts, Bellaire, Texas, United States

REFERENCES:
- [Result] Hemsen L, Cusack SL, Minkowitz HS, Kuss ME. A feasibility study to investigate the use of a bupivacaine-collagen implant (XaraColl) for postoperative analgesia following laparoscopic surgery. J Pain Res. 2013;6:79-85. doi: 10.2147/JPR.S40158. Epub 2013 Feb 1. PMID 23390367

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: Bupivacaine Collagen Sponge: 4, 5x5 bupivacaine collagen sponges
  4, 5x5cm bupivacaine collagen sponges
Period: Overall Study
Arm/Group | Drug: Bupivacaine Collagen Sponge
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Drug: Bupivacaine Collagen Sponge
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Use of Opioid Analgesia - Morphine Equivalence (mg)
Description: Dosages of 1 to 2 mg per dose were titrated to patient comfort according to institutional standards and at the investigator's discretion. Once patients could tolerate oral medication, they were offered oral morphine (15 mg tablets) as rescue analgesia if necessary. The dose for patients who weighed less than 75kg was 15mg every 3 to 4 hours as needed for pain control. The dose for patients who weighed 75kg or more was 1-2 tablets (15-30 mg) every 3-4 hours for pain control. Morphine was the preferred rescue medication.
Time Frame: 0 to 24 hours after surgery
Measure: Mean (Standard Deviation); unit: Morphine Equivalence (mg)
Groups:
- Bupivacaine Collagen Sponge: Bupivacaine Collagen Sponge
Arm/Group | Bupivacaine Collagen Sponge
Number analyzed (Participants) | 10
Morphine Equivalence (mg) | 19.3 (15.5)

2. Primary Outcome: Total Use of Opioid Rescue Analgesia - Morphine Equivalence (mg)
Description: as for outcome 1
Time Frame: 25-48 hours
Measure: Mean (Standard Deviation); unit: Morphine Equivalence (mg)
Groups:
- Bupivacaine Collagen Sponge: 4, 5x5 bupivacaine collagen sponges
Arm/Group | Bupivacaine Collagen Sponge
Number analyzed (Participants) | 10
Morphine Equivalence (mg) | 5.3 (7.3)

3. Primary Outcome: Total Use of Opioid Rescue Analgesia - Morphine Equivalence (mg)
Description: as for outcome 1
Time Frame: 49-72 Hours
Measure: Mean (Standard Deviation); unit: Morphine Equivalence (mg)
Arm/Group | Bupivacaine Collagen Sponge
Number analyzed (Participants) | 10
Morphine Equivalence (mg) | 2.0 (3.3)

4. Primary Outcome: Total Use of Opioid Rescue Analgesia Morphine Equivalence (mg)
Description: as for outcome 1
Time Frame: 0-48 hours)
Measure: Mean (Standard Deviation); unit: Morphine Equivalence (mg)
Arm/Group | Bupivacaine Collagen Sponge
Number analyzed (Participants) | 10
Morphine Equivalence (mg) | 24.6 (21.8)

5. Primary Outcome: Total Use of Opioid Rescue Analgesia - Morphine Equivalence (mg)
Description: as for outcome 1
Time Frame: 0-72 hours
Measure: Mean (Standard Deviation); unit: Morphine Equivalence (mg)
Arm/Group | Bupivacaine Collagen Sponge
Number analyzed (Participants) | 10
Morphine Equivalence (mg) | 26.6 (23.2)

ADVERSE EVENTS:
Groups:
- Drug: Bupivacaine Collagen Sponge: 4, 5x5 bupivacaine collagen sponges
Arm/Group | Drug: Bupivacaine Collagen Sponge
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: Bupivacaine Collagen Sponge (N=10)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: Bupivacaine Collagen Sponge (N=10)
Headache (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Scrotal Swelling (Reproductive system and breast disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Post-op Tremors (General disorders) | 1 (1)
Effusion at Hernia Site (General disorders) | 1 (1)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No